CLINICAL TRIAL: NCT06807177
Title: Can Blood Biomarkers of Inflammation and BDNF be Used to Assess the Effectiveness of Collagen Mesotherapy in Chronic Cervical Myofascial Pain Syndrome?
Brief Title: Can Blood Biomarkers of Inflammation and BDNF be Used to Assess the Effectiveness of Collagen Mesotherapy in Chronic CMPS?
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Responsible Party: Sponsor
Other Study IDs: KBT-517/2022
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain Syndrome - Neck; Spondyloarthrosis; Neck Pain; Cervical Pain
Keywords: mesotherapy; tnf alpha; interleukin 6; collagen type I; lignocaine; interleukin 1-beta
MeSH Terms: conditions — Spondylarthritis; Neck Pain; Osteogenesis Imperfecta, Type IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be collected as serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Injection type I collagen
- Injection 1% lignocaine

SUMMARY:
The aim of the study is to assess the concentration of anti-inflammatory markers after the use of cervical spine mesotherapy in the course of pain syndrome. The study is randomized. Patients will be divided into two groups: A - mesotherapy using injectable type I collagen, B - mesotherapy using 1% lignocaine. The mesotherapy procedure will be performed five times, at weekly intervals. Blood will be collected before the start of mesotherapy, a week after its completion and after 3 months of follow-up. In addition, the effectiveness and safety of mesotherapy of the cervical spine will be assessed.

DETAILED DESCRIPTION:
Study aim:

The main objective of this article was to answer the question: Can biomarkers of inflammatory processes in the blood and BDNF be used to evaluate the effectiveness of collagen mesotherapy in chronic CMPS? The second objective of this article is to evaluate the safety of collagen mesotherapy in chronic CMPS.

Material and methods:

The study was conducted on patients aged 18 to 80 years, of both sexes, with local, chronic cervical spine pain syndrome, without radiation of symptoms to the upper limb. The study subjects were recruited at the National Institute of Geriatric, Rheumatology and Rehabilitation in Warsaw. Patients will be recruited according to the inclusion and exclusion criteria. The study is randomized. Patients will be divided into two groups: A - mesotherapy using injectable type I collagen, B - mesotherapy using 1% lignocaine.

Each patient will have blood collected before starting mesotherapy (on the same day) to determine anti-inflammatory markers (TNF-alpha, interleukin-1-beta, interleukin-6) and BDNF. Again, a week after the end of mesotherapy (five treatments) and after 6-week of follow-up, blood will be collected to determine the same markers.

In addition, the effectiveness and safety of mesotherapy of the cervical spine will be assessed. A Numeric Rating Scale (VAS) and the Neck Disability Index (NDI) scale will be used.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic (>12 weeks) cervical spine pain syndrome of muscular, myofascial nature without radiation to the upper limb
* recent MRI or CT scan of the cervical spine (up to 6 months)
* no serious diseases: cancer, rheumatology, metabolic
* no allergy to lignocaine 1% or injectable type I collagen

Exclusion Criteria:

* another cause of cervical spine pain
* lack of patient consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic cervical spine pain, of a muscular, myofascial and overload nature, will be qualified for the study and undergo spinal mesotherapy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of anti-inflammatory markers | Blood collection before starting the mesotherapy treatment (on the same day), one week after its completion (after 5 weeks from start), and after 6 weeks from end
  Blood collection before starting the mesotherapy treatment (on the same day), one week after its completion, and after 6 weeks follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Geriatric, Rheumatology and Rehabilitation, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No